CLINICAL TRIAL: NCT04914065
Title: Predictors of Prognosis in Patients With Critical Illness.
Status: Completed | Type: Observational
Sponsor: Taoyuan General Hospital (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other); Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: TYGH108031
Record Dates: First submitted 2021-05-25; First posted 2021-06-04 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: ICU Acquired Weakness; Weaning Failure; Quality of Life
Keywords: Intensive care unit acquired weakness; Handgrip strength; Muscle thickness; Predictor; Ventilator weaning; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Regular care in the surgery intensive care unit — Part 1: Two arms(muscle thickness observation):
  1. Inspiratory muscles: diaphragm
  2. Anti-gravity muscles: rectus femoris and the vastus intermedius
  Part 2: Predictors of short-term and long-term goals in the ICU
  1. Short-term goal: successful ventilator weaning in the ICU- pass weaning profile without re-intubation in the hospital
  2. Long-term goal- Quality of life after hospital discharge: SF-36 (Taiwan version)

SUMMARY:
Recently, intensive care unit acquired weakness (ICUAW) has become a hotspot issue in the patients with critical illness. The symptoms of ICUAW, including sensory impairment and muscle atrophy, may lead to poor quality of life even though the patients discharged from the ICU for a long time. Therefore, an ounce of prevention is worth a pound of cure. At the same time, early evaluation is necessary to keep critically ill patients away from ICUAW. Medical Research Council (MRC) scale is the most common approach for diagnosis clinically. Regarding the interrater variation of MRC, handgrip strength (HGS) has been thought to be a simple and accurate alternative. However, HGS does not belong to antigravity or respiratory muscle which are the first to be affected by immobilization. It is still unknown whether HGS can represent the general muscle condition in ICU or not.

Additionally, previous studies have proved that patients with critical illness in the ICU would have better prognosis and less complications, if they undergo physical therapy as soon as possible. In addition to early ventilator weaning and reduced mortality rate, physical therapy could enhance quality of life (QoL) after patient discharges from hospital. However, early mobility in the ICU mainly emphasizes cardiopulmonary patients due to the traditional concept in Taiwan. Hence, the duration of mechanical ventilation in the critical patients will affect the timing to receive physical therapy, even impact the improvement of QoL.

Because of these reasons, this study will investigate the relationship between HGS and muscle mass among patients with critical illness and find the predictors of the short-term and long-term goals in the ICU, including ventilator weaning and QoL after hospital discharge.

DETAILED DESCRIPTION:
This prospective and observational study will be divided into 2 parts: 1) The association between handgrip strength and muscle mass in intensive care unit patients. 2) Predictors of short-term and long-term goals in ICU.

Patients in the surgery intensive care unit of Taoyuan General Hospital will be recruited and evaluated in 48 hours from admission to ICU. The outcome measures include HGS assessed by electronic hand dynamometer and muscle thickness of diaphragm and quadriceps detected by ultrasound.

The short-term goal is weaning ventilator, and the long-term goal is quality of life after discharge from hospital assessed through SF-36 Taiwan version. Patients in the surgery intensive care unit of Taoyuan General Hospital will be recruited and evaluated in 48 hours after ICU admission. The collected data contain muscle strength, muscle mass, physical function, respiratory function, and observation of delirium or not. The evaluations of muscle strength include 3 parts which are limbs(handgrip), respiratory muscle(Maximal Inspiratory Pressure), and general muscle strength(Medical Research Council scale); Secondly, the evaluations of muscle mass divide 2 parts which are limbs(muscle thickness of quadriceps) and respiratory muscle(muscle thickness of diaphragm); Thirdly, the evaluations of physical function are 2 ways which are FSS-ICU and 2 mins walk test after discharge from the ICU; Fourthly, the evaluations of respiratory function contain 3 measurements of FEV1, FVC, and FEV1/FVC; Finally, the evaluation of delirium is assessed by CAM-ICU.

The statistical analysis will use SPSS version 24. Pearson correlation test will be conducted to investigate the association between HGS and muscle thickness. Multiple regression will be used to investigate the predictors for weaning ventilator successfully and quality of life after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the surgery intensive care unit will be recruited and evaluated in 48 hours from admission to ICU

Exclusion Criteria:

* Hemodynamic instability patients, e.g., patients with ECMO
* Patients refuse to participate this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the surgery intensive care unit will be recruited and evaluated in 48 hours from admission to ICU
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Change of handgrip strength (HGS) from ICU admission to ICU discharge | every day during the ICU stay until patients discharge from ICU assessed up to 14 days
  Handgrip strength (HGS) assessed by electronic hand dynamometer(Electronic hand dynamometer, CAMRY, MODEL, EH101)
Part 1: Change of diaphragm thickness from ICU admission to ICU discharge | every day during the ICU stay until patients discharge from ICU assessed up to 14 days
  Muscle thickness of diaphragm and quadriceps detected by ultrasound(GE vivid S5)
Part 2: Change of Handgrip strength (HGS) | Baseline: admission to ICU in 48 hours. Progress: the day that patients received weaning profile test
  Change of Handgrip strength (HGS) assessed by electronic hand dynamometer(Electronic hand dynamometer, CAMRY, MODEL, EH101)
Part 2: Change of General muscle strength | Baseline: admission to ICU in 48 hours. Progress: the day that patients received weaning profile test
  Change of General muscle strength- MRC scale
Part 2: Change of Muscle mass | Baseline: admission to ICU in 48 hours. Progress: the day that patients received weaning profile test
  Muscle thickness of diaphragm and quadriceps detected by ultrasound (GE vivid S5)
Part 2: Respiratory muscle strength | the day that patient received weaning profile tests during ICU
  Respiratory muscle strength- Maximal Inspiratory Pressure(MIP)
Part 2: Change of Physical function | Baseline: admission to ICU in 48 hours. Progress: the day that patients received weaning profile test
  Change of FSS-ICU
Part 2: Physical function at ICU discharge | conducted at the day of ICU discharge
  2 mins walk test
Part 2: Change of Delirium | conducted every day in the ICU
  CAM-ICU
Part 2: Respiratory function | conducted at the day of ICU discharge
  FVC, FEV1, FEV1/ FVC assessed by ezOxygen (EZO-G001)
Part 2: Quality of life- SF-36(Taiwan version) | conducted by phone call at discharge for 6 months from ICU
  SF-36(Taiwan version)

CONTACTS AND LOCATIONS:
Overall Officials: Huan-Jui Yeh, Study Chair — Department of Rehabilitation, Taoyuan General Hospital, Ministry of Health and Welfare
Locations (1):
- Department of Rehabilitation, Taoyuan General Hospital, Ministry of Health and Welfare, Taiwan, Taoyuan District, Taiwan

REFERENCES:
- [Background] Thille AW, Boissier F, Muller M, Levrat A, Bourdin G, Rosselli S, Frat JP, Coudroy R, Vivier E. Role of ICU-acquired weakness on extubation outcome among patients at high risk of reintubation. Crit Care. 2020 Mar 12;24(1):86. doi: 10.1186/s13054-020-2807-9. PMID 32164739
- [Background] Meyer-Friessem CH, Malewicz NM, Rath S, Ebel M, Kaisler M, Tegenthoff M, Schildhauer TA, Pogatzki-Zahn EM, Maier C, Zahn PK. Incidence, Time Course and Influence on Quality of Life of Intensive Care Unit-Acquired Weakness Symptoms in Long-Term Intensive Care Survivors. J Intensive Care Med. 2021 Nov;36(11):1313-1322. doi: 10.1177/0885066620949178. Epub 2020 Aug 17. PMID 32799703
- [Background] Cottereau G, Dres M, Avenel A, Fichet J, Jacobs FM, Prat D, Hamzaoui O, Richard C, Antonello M, Sztrymf B. Handgrip Strength Predicts Difficult Weaning But Not Extubation Failure in Mechanically Ventilated Subjects. Respir Care. 2015 Aug;60(8):1097-104. doi: 10.4187/respcare.03604. Epub 2015 Mar 10. PMID 25759461
- [Background] Kutchak FM, Rieder MM, Victorino JA, Meneguzzi C, Poersch K, Forgiarini LA Junior, Bianchin MM. Simple motor tasks independently predict extubation failure in critically ill neurological patients. J Bras Pneumol. 2017 May-Jun;43(3):183-189. doi: 10.1590/S1806-37562016000000155. PMID 28746528
- [Background] Saiphoklang N, Tepwimonpetkun C. Interest of hand grip strength to predict outcome in mechanically ventilated patients. Heart Lung. 2020 Sep-Oct;49(5):637-640. doi: 10.1016/j.hrtlng.2020.03.019. Epub 2020 May 6. PMID 32387152
- [Background] Braganca RD, Ravetti CG, Barreto L, Ataide TBLS, Carneiro RM, Teixeira AL, Nobre V. Use of handgrip dynamometry for diagnosis and prognosis assessment of intensive care unit acquired weakness: A prospective study. Heart Lung. 2019 Nov-Dec;48(6):532-537. doi: 10.1016/j.hrtlng.2019.07.001. Epub 2019 Jul 15. PMID 31320179
- [Background] Jolley SE, Bunnell AE, Hough CL. ICU-Acquired Weakness. Chest. 2016 Nov;150(5):1129-1140. doi: 10.1016/j.chest.2016.03.045. Epub 2016 Apr 7. PMID 27063347
- [Background] Sidiras G, Patsaki I, Karatzanos E, Dakoutrou M, Kouvarakos A, Mitsiou G, Routsi C, Stranjalis G, Nanas S, Gerovasili V. Long term follow-up of quality of life and functional ability in patients with ICU acquired Weakness - A post hoc analysis. J Crit Care. 2019 Oct;53:223-230. doi: 10.1016/j.jcrc.2019.06.022. Epub 2019 Jun 21. PMID 31277049
- [Background] Supinski GS, Morris PE, Dhar S, Callahan LA. Diaphragm Dysfunction in Critical Illness. Chest. 2018 Apr;153(4):1040-1051. doi: 10.1016/j.chest.2017.08.1157. Epub 2017 Sep 5. PMID 28887062
- [Background] Vanhorebeek I, Latronico N, Van den Berghe G. ICU-acquired weakness. Intensive Care Med. 2020 Apr;46(4):637-653. doi: 10.1007/s00134-020-05944-4. Epub 2020 Feb 19. PMID 32076765
- [Background] Bohannon RW, Wang YC, Gershon RC. Two-minute walk test performance by adults 18 to 85 years: normative values, reliability, and responsiveness. Arch Phys Med Rehabil. 2015 Mar;96(3):472-7. doi: 10.1016/j.apmr.2014.10.006. Epub 2014 Oct 25. PMID 25450135
- [Background] Fuke R, Hifumi T, Kondo Y, Hatakeyama J, Takei T, Yamakawa K, Inoue S, Nishida O. Early rehabilitation to prevent postintensive care syndrome in patients with critical illness: a systematic review and meta-analysis. BMJ Open. 2018 May 5;8(5):e019998. doi: 10.1136/bmjopen-2017-019998. PMID 29730622
- [Background] Zein H, Baratloo A, Negida A, Safari S. Ventilator Weaning and Spontaneous Breathing Trials; an Educational Review. Emerg (Tehran). 2016 Spring;4(2):65-71. PMID 27274515